CLINICAL TRIAL: NCT03186391
Title: Sensitivity and Specificity of the AHA Post-exercise ABI Criteria
Brief Title: Exercise Testing in Peripheral Artery Disease Patients
Acronym: ExercisePAD
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_3064
Record Dates: First submitted 2017-05-23; First posted 2017-06-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected PAD: Use the data collected during a usual consultation to study the relationship between different parameters (rest pressure ...) and imaging
  Interventions: Other: Data collected

INTERVENTIONS:
Other: Data collected — Use the data collected during a usual consultation to study the relationship between different parameters (rest pressure ...) and imaging

SUMMARY:
The aim of this study was to evaluate exercise testing in case of patients suspected of Peripheral Artery Disease (PAD).

DETAILED DESCRIPTION:
This is a non interventional prospective cross sectional, monocentric study. All patients addressed in our vascular unit for exercise testing were included. All patients' data performed in clinical routine can be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients addressed in our vascular unit for exercise limitation

Exclusion Criteria:

* Incapacity to walk on the treadmill.
* A severe cardiopathy contraindicating a stress test

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to our vascular unit with exercise limitation
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2014-02-24 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
1-min Post-exercise Ankle-Brachial Index (ABI) | at 1 minute after the stop of walking
  Post exercise pressures at 1 minute after the stop of walking on each ankle and arm.

SECONDARY OUTCOMES:
3-min Post-exercise Ankle-Brachial Index (ABI) | at 3 minutes after the stop of walking
  Post exercise pressures at 3 minutes after the stop of walking on each ankle and arm.
5-min Post-exercise Ankle-Brachial Index (ABI) | at 5 minutes after the stop of walking
  Post exercise pressures at 5 minutes after the stop of walking on each ankle and arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mahé Guillaume, MD-PhD, Principal Investigator — Rennes University Hospital
Locations (1):
- Centre hospitalier Universitaire, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vannier C, Guezais A, Talbot M, Le Faucheur A, Mahe G. Relationship between exercise transcutaneous oxygen pressure measurements with constant and graded treadmill tests. Vasc Med. 2025 Dec;30(6):676-682. doi: 10.1177/1358863X251379810. Epub 2025 Nov 5. PMID 41193436
- [Derived] Metairie A, Tollenaere Q, Laneelle D, Le Faucheur A, Le Pabic E, Omarjee L, Mahe G. Simplification of ankle-brachial-index measurement using Doppler-waveform classification in symptomatic patients suspected of lower extremity artery disease. Front Cardiovasc Med. 2022 Sep 9;9:941600. doi: 10.3389/fcvm.2022.941600. eCollection 2022. PMID 36158813